CLINICAL TRIAL: NCT05638672
Title: A Multicenter, Double-blind, Double-dummy, Randomized, Parallel-controlled Clinical Study Evaluating Huashi Baidu Formula in the Treatment of Mild and Moderate Types of COVID-19 Disease.
Brief Title: COVID-19 Huashi Baidu Formula Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Beijing YouAn Hospital (Other); Kossamak Hospital (Unknown); Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022XLA151-2
Record Dates: First submitted 2022-12-05; First posted 2022-12-06 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: Huashi Baidu Granule; Randomized controlled trial; Evidence-based
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Huashi Baidu Granule+Monapiravir simulant
  Interventions: Drug: Huashi Baidu Granule
- Control group (Active Comparator): Monapiravir+Huashi Baidu Granule Simulator
  Interventions: Drug: Monapiravir

INTERVENTIONS:
Drug: Huashi Baidu Granule — Granule is produced by Guangdong Yifang Pharmaceutical Co., Ltd. with a specification of 5g × 12 bags, twice a day, take 2 sachets each time with boiling water.
  Arms: Treatment group
Drug: Monapiravir — Monapiravir, manufactured by Merck, an American pharmaceutical company, with the specification of 200mg × 40 capsules, 800mg each time, twice a day.
  Arms: Control group

SUMMARY:
Combined with the regional and population characteristics of Asia and Africa, Huashi Baidu Granule was used to intervene in mild and moderate patients with COVID-19, evaluate its efficacy and safety, and clarify its characteristics of action.

DETAILED DESCRIPTION:
In this study, a double-blind, double dummy, randomized control method was used to include 300 cases of mild and moderate COVID-19 patients in three centers at home and abroad. The clinical efficacy of Huashi Baidu Granule and Monapiravir in intervening COVID-19 patients was compared, It is proved that Huashi Baidu Granule has the same clinical efficacy and safety against COVID-19 as Monapiravir, and its characteristics of action are clarified to obtain high-level clinical evidence-based medical evidence of Huashi Baidu Granule in treating COVID-19 mild and moderate.

ELIGIBILITY:
Inclusion Criteria:

1. Conform to the diagnostic criteria for COVID-19 mild and moderate in the Guidelines for the Diagnosis and Treatment of Novel Coronavirus (COVID-19) Infection (Trial Version 10) ；
2. Age ≥ 18 years and ≤ 65 years;
3. The time from the first symptom (or confirmed onset) shall not exceed 5 days;
4. If the patient agrees to participate in the study, he/she will sign the informed consent form through paper signature, electronic signature of mobile software or voice authorization.

Exclusion Criteria:

1. Patients who cannot guarantee the compliance of taking medicine during the treatment period, and who are difficult to take medicine by oral or nasal feeding.
2. Patients with severe primary respiratory diseases or other pathogenic microorganism pneumonia that needs to be differentiated from COVID-19.
3. Pregnant women, with positive urine pregnancy test, or with pregnancy plan within 12 months.
4. Patients suffering from malignant tumors, mental diseases and other systematic malignant diseases that the researchers consider unsuitable for the study.
5. People who have ever been allergic to the test drug and who do not tolerate the drug.
6. Those who are participating in other clinical trials.
7. Non severe patients in the trial shall not enter the study again after changing the classification.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-06 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Nucleic acid negative rate in 5 days;Virus CT value | The treatment period，Receive the test by PCR once a daily ，for 5 consecutive days
  Quantitative standard of viral CT value for nucleic acid detection： According to the Technical guidelines for laboratory testing of novel coronavirus, the Ct value of nucleic acid testing of novel coronavirus is less than 37, which can be reported is positive; No Ct value or Ct value greater than 40 was negative. If the Ct value was between 37 and 40, it is recommended to repeat the experiment. If Ct If the value is less than 40, the amplification curve has obvious peak, and the sample is judged as positive, otherwise it is negative.

SECONDARY OUTCOMES:
Disease score | The treatment period, including 5 days after administration, and the follow-up period, which is day 11, day 21, and day 30 after administration, respectively
  Therapeutic efficacy evaluation scale of traditional Chinese medicine in treating COVID-19
Score of individual symptom | The treatment period, including 5 days after administration, and the follow-up period, which is day 11, day 21, and day 30 after administration, respectively
  fever, asthenia, cough, dyspnea, generalized aches and pains, abnormal taste and smell, diarrhea, nasal congestion, runny nose and headache
TCM symptom score | The treatment period, including 5 days after administration, and the follow-up period, which is day 11, day 21, and day 30 after administration, respectively
  Quantitative table of TCM syndrome score of novel coronavirus pneumonia
Hematological parameters | The treatment period, day one and day five after administration
  C-reactive protein, erythrocyte sedimentation rate, lymphocyte count, lymphocyte/neutrophil ratio, coagulation, D-Di and IL-6
Symptom relief rate | 30days
  Time when symptom disappears
Rate of progression to severe COVID-19 cases | 30days
  Refer to the severe diagnostic criteria for COVID-19 issued by the National Health Commission and the National Administration of Traditional Chinese Medicine: Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing You'an Hospital, Capital Medical University, Beijing, Beijing Municipality, China